CLINICAL TRIAL: NCT05037903
Title: Cognitive-Behavioral Therapy for Adults With Attention-Deficit/Hyperactivity Disorder Inattentive Presentation: A Qualitative Study
Brief Title: Cognitive-Behavioral Therapy for Adults With ADHD: A Qualitative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Benjamin Bohman, Study Principal Investigator, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KI-2021-01663
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive-behavioral therapy (Experimental): Cognitive-behavioral therapy, including behavioral exercises and homework assignments.
  Interventions: Behavioral: Cognitive-behavioral therapy

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy — Cognitive and behavioral interventions aimed at increasing behavioral activation, and reducing procrastination and inattentive symptoms.

SUMMARY:
This is a qualitative study of participants who have taken part in a randomized controlled trial (RCT) of a new treatment protocol based on cognitive-behavioral therapy for adults with attention deficit/hyperactivity disorder predominantly inattentive presentation. The purpose of the qualitative study is to explore participant perceptions of taking part in the RCT to further develop and improve the new treatment protocol.

ELIGIBILITY:
Inclusion Criteria:

* Principal diagnosis of ADHD inattentive presentation
* 18 years of age or older
* If on medication, it needs to be well-established since three months, and
* Prior psycho-educational intervention

Exclusion Criteria:

* Intellectual impairment
* Substance use disorder
* Difficulties in adherence to medical or other treatment
* Social and/or psychiatric problems to such an extent that they prevent focusing on treatment, or
* Simultaneous psychological treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Qualitative interview data | 45-60 minutes
  Participant responses based on questions posed in an interview

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Bohman, Principal Investigator — Karolinska Institutet
Locations (1):
- Stockholm Health Care Services, Region Stockholm, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stralin EE, Sunnhed R, Thorell LB, Lundgren T, Bolte S, Bohman B. "It was very nice to be in a room where everyone had ADD-that's kind of VIP": Exploring clients' perceptions of group CBT for ADHD inattentive presentation. PLoS One. 2024 Jun 21;19(6):e0299060. doi: 10.1371/journal.pone.0299060. eCollection 2024. PMID 38905212